CLINICAL TRIAL: NCT00665535
Title: Preventing Pressure Ulcers: A Multi-site RCT in Nursing Facilities
Brief Title: Pressure Ulcer Prevention: Turning for Ulcer Reduction
Acronym: TURN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH); National Institute on Aging (NIA) (NIH); Ontario Ministry of Health and Long Term Care (Other Government); Toronto Health Economic Technology Assessment collaborative (THETA) (Unknown)
Responsible Party: Principal Investigator, Nancy Bergstrom, Trumble Professor of Aging Research & Director, Center on Aging, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R011NR009680-01A1
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; Nursing facilities; Elderly; At risk for pressure ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2. High Risk (Other): High risk for pressure ulcers according to the Braden Scale for Predicting Pressure Sore Risk (Score 10-12)
  Interventions: Procedure: Turning or repositioning schedule
- 1. Moderate Risk (Other): Moderate risk for pressure ulcers according to the Braden Scale for Predicting Pressure Sore Risk (Score 13 and 14)
  Interventions: Procedure: Turning or repositioning schedule

INTERVENTIONS:
Procedure: Turning or repositioning schedule — Turning schedule randomly assigned at 2, 3, or 4 hours
  Arms: 1. Moderate Risk
Procedure: Turning or repositioning schedule — Turning schedule randomly assigned at 2, 3 or 4 hours
  Arms: 2. High Risk

SUMMARY:
The purpose of the study is to determine the optimal frequency of repositioning nursing facility residents with limited mobility who are cared for on a high density foam mattress in order to prevent bed sores. It is hypothesized that participants at moderate risk (Braden Scale Scores 13-14) who are turned every 3 or 4 hours and participants at high risk (Braden Scores 10-12) turned every 3 or 4 hours will not have a higher incidence of ulcers than those residents turned every 2 hours.

DETAILED DESCRIPTION:
The purpose of this multi-site, randomized, controlled trial is to determine the optimal frequency of repositioning nursing facility residents with mobility limitations who are at moderate and high risk for pressure ulcer development who are cared for on high density foam mattresses for the purpose of preventing pressure ulcers. Pressure ulcers result primarily from pressure over a bony prominence that occludes blood flow to tissues. Traditionally, soft surfaces over mattress and repositioning individuals every 2 hours to relieve pressure have been the gold standard of care to prevent ulcers. Recent improvements in support surfaces may reduce the need for 2-hour repositioning. The specific aims of this study are to determine if: 1) there is a significant difference in the incidence of pressure ulcers among: a) moderate risk (Braden Scale Score, 13-14) residents randomly assigned to be repositioned every 2-, compared with every 3- or 4- hours; or b) high risk (Braden Scale Score, 10-12) residents who are turned every 2- compared with every 3- or 4-hours; 2) mobility (spontaneous or assisted) measured by actigraphy is a significant covariate with repositioning frequency in the incidence of pressure ulcers and 3) resident characteristics and resident influencing factors are significant covariates of repositioning schedules on pressure ulcer incidence. A 2 X 2/2 X 3 experimental design is used in which participants at two levels of risk (moderate or high) for pressure ulcer development are randomly assigned to one of 3 repositioning schedules every 2-hours (the current standard of care), contrasted with 3- or 4- hours carried out for 3 weeks. Actigraphs worn for 7 days (Tuesday to Tuesday) will determine if mobility is a significant covariate. Residents (1080) who are over 65 years, able to give consent or have a surrogate who can give consent and are at moderate or high risk for pressure ulcers will be invited to participate. Nursing facilities are selected because of their ability to follow a research protocol and submit data according to protocol requirements, and who have a reputation for good care are being selected for participation. Participants will be randomly assigned to a repositioning schedule that will be carried out by a Certified Nursing Assistants (CNA) who will document time of each repositioning. A CNA supervisor monitors repositioning and documentation frequently. Data are FAXED to and monitored by the investigators daily. With the exception of the repositioning intervention, participants will receive the same preventive care as all residents. The primary outcome of this study, pressure ulcers (yes/no) will be documented by a nurse assessor who will be masked to the repositioning timing. Data analysis and management will be performed by ISIS. The goal of this study is to shape Nursing Facility policy by defining how level of risk, mobility, and frequency of repositioning of residents can reduce the incidence of pressure ulcers and improve resident outcomes. Less frequent repositioning would allow residents longer periods of sleep, would reduce staff time for repositioning, and allow more efficient allocation of time.

ELIGIBILITY:
Inclusion Criteria: Participants will:

* Be free of pressure ulcers upon admission to the study.
* Have a Braden Scale Score between 10 - 12 (high risk) or 13 -14 (moderate risk) within one week of admission (new residents) or greater than 90 days (established residents) of study participation
* Have a high-density foam replacement mattress in use or can be transferred to such a mattress.
* Are 65 years or older. Younger residents are present in fewer numbers and may have different health issues and co-morbidities than older residents.
* Can legally grant consent to participate or have available surrogates to grant consent. If able, participant should assent when a surrogate grants consent.
* Expected to have a length of stay of 21 days or greater.

Exclusion Criteria:

* Pressure ulcer is present upon initial examination.
* The Braden Scale score is 15 or greater indicating mild risk or no risk, or 9 or below indicating very high risk.
* The resident cannot be turned on 3 anatomical surfaces (side, back, side) or has a contraindication to repositioning.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 967 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pressure ulcers, present (stage)or absent | End of 3rd week or conclusion of participation

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bergstrom, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Susan Horn, PhD, Principal Investigator — ISIS, Salt Lake City, UT
Locations (26):
- United States (19):
  - Glencroft Care Center, Glendale, Arizona
  - Linda Valley Nursing Facility, Loma Linda, California
  - Garden Crest Convalescent Hospital, Los Angeles, California
  - St. Catherine Laboure Manor, Jacksonville, Florida
  - Miami Jewish Home & Hospital, Miami, Florida
  - Palatka Health Care Center, Palatka, Florida
  - Kindred Bremen Health Care Center, Bremen, Indiana
  - Tower Hill Center for Health and Rehabilitation, Canton, Massachusetts
  - Gurwin Jewish Nursing and Rehabilitation Center, Commack, New York
  - Monroe Community Hospital, Rochester, New York
  - BlumenthalJewish Nursing and Rehabilitation, Greensboro, North Carolina
  - Hennis Care Center, Dover, Ohio
  - Dorothy Love Retirement Community, Sidney, Ohio
  - Fairmount at aBreckenridge Village, Willoughby, Ohio
  - Park Vista Retirement Community, Youngstown, Ohio
  - Signature HealthCare of Columbia, Columbia, Tennessee
  - Kindred Loudon Healthcare Center, Loudon, Tennessee
  - Kindred Fairpark Health Care Center, Maryville, Tennessee
  - Asbury Place Maryville, Maryville, Tennessee
- Canada (7):
  - Tyndall Nursing Home, East Missassauga, Ontario
  - Malton Village Long Term Care Center, Mississauga, Ontario
  - Specialty Care of Mississauga Road, Mississauga, Ontario
  - Yee Hong Scarborough, Scarborough Village, Ontario
  - Shepherd Lodge, Scarborough Village, Ontario
  - Leisure World Lawrence, Toronto, Ontario
  - Villa Leonardo Gambin Specialty Care, Woodbridge, Ontario

REFERENCES:
- [Derived] Yap TL, Kennerly SM, Bergstrom N, Hudak SL, Horn SD. An Evidence-Based Cue-Selection Guide and Logic Model to Improve Pressure Ulcer Prevention in Long-term Care. J Nurs Care Qual. 2016 Jan-Mar;31(1):75-83. doi: 10.1097/NCQ.0000000000000128. PMID 26066791
- [Derived] Omolayo T, Brown K, Rapp MP, Li J, Barrett R, Horn S, Bergstrom N. Construct validity of the moisture subscale of the Braden Scale for Predicting Pressure Sore Risk. Adv Skin Wound Care. 2013 Mar;26(3):122-7. doi: 10.1097/01.ASW.0000427921.74379.c5. PMID 23426413
- See also: Home of the Braden Scale and source of official copies of the tool and the location for obtaining permission to use the tool. — http://www.bradenscale.com
- See also: Home of the National Pressure Ulcer Advisory Panel with information regarding staging and policies regarding pressure ulcers — http://www.npuap.org/
- See also: Home page of the Wound Ostomy and Continence Nurses Organization, the experts in wound healing. — http://www.wocn.org/
- See also: Hennis Care Center of Dover, Ohio is a data collection site — http://www.henniscarecentre.com/volunteers.htm
- See also: Gurwin Jewish Nursing and Rehabilitation Center, Commack, NY, is a data collection site — http://www.gurwin.org/
- See also: Monro Community Hospital, Rochester, NY, is a data collection sites — http://www.monroehosp.org/
- See also: Specialty Care Mississauga Road, Mississauga, Ontario, Canada is a data collection site — http://www.specialty-care.com/index.php/mississauga-road
- See also: Villa Leonardo Gambin, Woodbridge, Ontario, Canada is a data collection site — http://www.specialty-care.com/index.php/villa-leonardo-gambin
- See also: Fairmount at Breckenridge Village is a data collection site — http://www.oprs.org/breckenridge_village/
- See also: St. Catherine Laboure Manor is a data collection site — http://www.jaxhealth.com/AboutUs/default.asp?ENOrgID=B8AD2776B8C74351ABCD7349B0C8D30D
- See also: Kindred Bremen Health Care Center — http://www.bremenhealthcare.com/BuildPageC.asp?IFacID=156&PageID=H
- See also: Miami Jewish Home & Hospital will be a data collection site — http://www.miamijewishhealthsystems.org
- See also: Kindred Fairpark Health Care Center is a data collection site — http://www.fairparkhc.com/BuildPageC.asp?IFacID=77&PageID=H
- See also: Kindred Loudon Healthcare Center is a data collection site — http://www.loudonhealthcare.com/BuildPageC.asp?IFacID=80&PageID=H
- See also: Related Info — http://www.bremenhealthcare.com
- See also: Related Info — http://www.miamijewishhealthsystems.org/
- See also: Related Info — http://www.signaturehealthcarellc.com/Facility/FacilityInfo.aspx